CLINICAL TRIAL: NCT02282878
Title: The Effect of Dietary Salt Intake on Immune Function in Patients With Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1406014201
Record Dates: First submitted 2014-10-31; First posted 2014-11-05 (Estimated); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Multiple Sclerosis
Keywords: High Sodium Diet; Low Sodium Diet; MS
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High/Low Sodium Diet (Experimental): All MS patients will receive 2 weeks of controlled high sodium diet followed by a 1 week washout and 2 weeks of low sodium diet.
  Interventions: Dietary Supplement: High/Low Sodium Diet
- High/Low Sodium Diet Control (Active Comparator): Age matched controls will receive two weeks of controlled high sodium diet followed by a 1 week washout and 2 weeks of low sodium diet.
  Interventions: Dietary Supplement: High/Low Sodium Diet

INTERVENTIONS:
Dietary Supplement: High/Low Sodium Diet — All patients will receive 2 weeks of the high sodium diet followed by a 1 week washout and then 2 weeks of the low sodium diet

SUMMARY:
The purpose of this work is to investigate the influence of dietary salt intake on immune function in multiple sclerosis (MS) subjects and healthy controls. This study primarily tests the hypothesis that higher dietary salt intake will be associated with a higher frequency of pathogenic Th17 cells and impaired function of protective regulatory T cells. If a relationship between dietary salt intake and immune function is observed, this study will also test: a) whether this relationship is unique to MS subjects or whether it is also present in healthy controls, and b) whether healthier immune function can be restored by restricting dietary salt intake.

DETAILED DESCRIPTION:
The purpose of this work is to investigate the influence of dietary salt intake on immune function in MS subjects and healthy controls. This study primarily tests the hypothesis that higher dietary salt intake will be associated with a higher frequency of pathogenic Th17 cells and impaired function of protective regulatory T cells. If a relationship between dietary salt intake and immune function is observed, this study will also test: a) whether this relationship is unique to MS subjects or whether it is also present in healthy controls, and b) whether healthier immune function can be restored by restricting dietary salt intake. This is a 5-week pilot study of a dietary intervention of 25 subjects with MS or Clinically Isolated Syndrome (CIS) by 2010 Diagnostic Criteria who will be identified and recruited from the Yale MS Center and/or referred from outside MS centers. 25 age-matched healthy controls will be recruited from friends, family members, spouses and the patient waiting room at the Yale MS Center.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female adult subjects
* Ages 18-60, inclusive
* diagnosis of CIS or MS by 2010 McDonald Criteria (in the case of MS subjects)
* Naive to FDA- approved MS therapies such as glatiramer acetate, interferon-beta, natalizumab, fingolimod, tecfidera, or teriflunomide

Exclusion Criteria:

* Secondary or primary progressive MS
* Prior exposure to FDA-approved MS therapies or chemotherapies of any kind
* Known history of autoimmune disease besides MS
* Known history of renal disease, hypertension or congestive heart failure
* Currently taking medications that could affect urine sodium excretion (e.g. diuretics or others that act on the renin-angiotensins-aldosterone system)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2014-09; Primary Completion 2018-12-19 (Actual); Study Completion 2019-12-08 (Actual)

PRIMARY OUTCOMES:
Number of Th17 cells | Change from baseline at 2 weeks
  Frequency of Th17 cells will be measured by flow cytometry through blood samples taken before and after each of the two week low sodium and high sodium diets

SECONDARY OUTCOMES:
Regulatory T cell function | Change from baseline at 2 weeks
  Frequency of regulatory T cells as measured by flow cytometry through blood samples taken before and after each of the two week low sodium and high sodium diets

CONTACTS AND LOCATIONS:
Overall Officials: David Hafler, MD, Principal Investigator — Yale University
Locations (1):
- Yale MS Center, New Haven, Connecticut, United States